CLINICAL TRIAL: NCT03710096
Title: Comparison of McGrath and Macintosh Laryngoscopes for Insertion of a Double Lumen Tube by Residents
Acronym: MacGrathDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017_65; 2018-A00789-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-10; First posted 2018-10-17 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Thoracic Injuries
Keywords: Mac Grath; Double lumen tube
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mac grath group (Experimental)
  Interventions: Device: macGrath
- Macintosh Group (Active Comparator)
  Interventions: Device: Macintosh's

INTERVENTIONS:
Device: macGrath — in the mac grath group we use the videolaryngoscope macGrath as first-line for the insertion of double lumen tube
  Arms: Mac grath group
Device: Macintosh's — in the macintosh group we use the laryngoscope with Macintosh's blade as first-line for the insertion of double lumen tube
  Arms: Macintosh Group

SUMMARY:
The insertion of double lumen tube is difficult even more if it is a resident with no experience. we think that using videolaryngoscopes for novice ones would facilitate insertion of double lumen tube thanks to the visualization on a LCD screen of the laryngeal structure.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic Surgery
* Insertion of double lumen tube

Exclusion Criteria:

* Emergency surgery
* Risk of inhalation
* Person unable to consent
* Persons deprived of liberty, under guardianship or trusteeship
* Pregnant or lactating woman
* Allergy to Tracrium, Propofol, Sufentanil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-11-04 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Rate of success of intubation in both groups at the first attempt | Baseline: one session
  the success is defined as a correct implementation of the probe endotracheal in double light by an internal of anesthesia in the 1st attempt.

SECONDARY OUTCOMES:
Individual Determination of Cormack Stage | Baseline: one session
  scoring system for the grading of direct laryngoscopy in case of tracheal intubation is difficult
Rate of good positioning of double lumen tube confirmed by fibroscopy | Baseline: one session
The rate of patients with an increase in systolic blood pressure of more than 20% compared to the measurement before insertion of the probe | Baseline: one session
Intubation time | Baseline: one session
The rate of patients with pharyngeal pains upon awakening | Baseline: one session

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Desbordes, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France